CLINICAL TRIAL: NCT06323382
Title: Efficacy of Locoregional Therapy Combined With Bevacizumab and PD1/L1 Inhibitor in Advanced Hepatocellular Carcinoma: a Multicenter, Observational, Real-world Study
Brief Title: Locoregional Therapy Combined With Bevacizumab and PD1/L1 Inhibitor in Advanced Hepatocellular Carcinoma
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhou Qunfang, Clinical Professor, Sun Yat-sen University
Other Study IDs: Liver Project 6
Record Dates: First submitted 2024-03-15; First posted 2024-03-21 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Advanced Hepatocellular Carcinoma; Anti-PD1/PDL1 Antibody; Bevacizumab
Keywords: Bevacizumab; Atezolizumab; Tislelizumab; Toripalimab; Sintilimab; Camrelizumab
MeSH Terms: interventions — Bevacizumab; atezolizumab; tislelizumab; toripalimab; sintilimab; camrelizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Locoregional therapy — TACE procedure The decision to utilize transarterial artery chemoembolization (TACE) was performed through the tumor-feeding artery. The embolization emulsion was a mixture of Epirubicin 30-60 mg, Lobaplatin 30-50 mg, and Lipiodol 10-30 ml, and it was infused into tumor-feeding arteries via a 2.7/2.8 Fr micro-catheter.
  HAIC procedure Hepatic arterial infusion chemotherapy (HAIC) procedure was performed with FOLFOX regimen: 85 or 135 mg/m2 oxaliplatin from hour 0 to 2 on day 1400 mg/m2 leucovorin from hour 2 to 4 on day 1, and 400 mg/m2 fluorouracil bolus at hour 5 on the day 1; and 2400 mg/m2 fluorouracil over 46 h on days 1 and 2.
  Other Names: TACE/HAIC
Drug: Bevacizumab — 15mg/kg or 7.5mg/kg intravenously every 3 weeks
Drug: Atezolizumab — 1200mg intravenously every 3 weeks
Drug: Tislelizumab — 200mg intravenously every 3 weeks
Drug: Toripalimab — 220mg intravenously every 3 weeks
Drug: Sintilimab — 200mg intravenously every 3 weeks
Drug: Camrelizumab — 200mg intravenously every 3 weeks

SUMMARY:
Atezolizumab + Bevacizumab was superior to sorafenib in overall survival in advanced hepatocellular carcinoma. The programmed cell death protein-1 (PD1) and PDL1 inhibitor, was effective and tolerable in patients with advanced hepatocellular carcinoma. We aimed to describe the efficacy and safety of locoregional therapy combined with Bevacizumab and PD1/L1 inhibitor in patients with advanced hepatocellular carcinoma who can not receive radical therapy.

DETAILED DESCRIPTION:
This study is a multicenter, observational real-world study to explore the efficacy, safety of locoregional therapy combined with Bevacizumab and PD1/L1 inhibitor in advanced hepatocellular carcinoma. This study focused on the management of locoregional therapy combined with Bevacizumab and PD-1/L1 inhibitor. This study will create a database that will provide clinical parameters and outcomes of patients undergoing locoregional therapy combined Bevacizumab and PD-1/L1 inhibitor as standard of care in hopes of answering key clinical questions.

ELIGIBILITY:
Inclusion Criteria:

1. HCC diagnosed by histopathological examination or Guidelines for Diagnosis and Treatment of Primary Liver Cancer or the recurrent HCC after surgery;
2. age between 18 and 75 years;
3. Stage B (middle stage) or C (late stage) HCC determined in accordance with Barcelona Clinic Liver Cancer staging system (BCLC stage).
4. Locoregional therapy include TACE or HAIC, locoregional combined with Bevacizumab and PD1/L1 inhibitor as firstline therapy; non-firstline therapy (previous use of any systemic therapy but intolerant or drug resistant).
5. Child-Pugh class A or B;
6. Eastern Cooperative Group performance status (ECOG) score of 0-2;
7. Hemoglobin ≥ 8.5 g/dL Total bilirubin ≤ 30mmol/L Serum albumin ≥ 32 g/L ASL and AST ≤ 5 x upper limit of normal Serum creatinine ≤ 1.5 x upper limit of normal INR ≤ 1.5 or PT/APTT within normal limits Absolute neutrophil count (ANC) >1,500/mm3
8. Prothrombin time ≤18s or international normalized ratio < 1.7.
9. Ability to understand the protocol and to agree to and sign a written informed consent document.

Exclusion Criteria:

1. Cholangiocellular carcinoma (ICC).
2. Patients without image information should be excluded;
3. The survival or patients less than 3 months.
4. Serious medical comorbidities.
5. Evidence of hepatic decompensation including ascites, gastrointestinal bleeding or hepatic encephalopathy.
6. Known history of HIV.
7. History of organ allograft.
8. Known or suspected allergy to the investigational agents or any agent given in association with this trial.
9. Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy.
10. Evidence of bleeding diathesis.
11. Patients with clinically significant gastrointestinal bleeding within 30 days prior to study entry.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study is a multicenter, observational real-world study to explore the efficacy, safety of locoregional therapy combined with Bevacizumab and PD1/L1 inhibitor in advanced hepatocellular carcinoma. This study focused on the management of locoregional therapy combined with Bevacizumab and PD-1/L1 inhibitor. This study will create a database that will provide clinical parameters and outcomes of patients undergoing locoregional therapy combined Bevacizumab and PD-1/L1 inhibitor as standard of care in hopes of answering key clinical questions.
Sampling Method: Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Progression-Free-Survival (PFS) | 12 months
  Progression was defined as progressive disease by independent radiologic review

SECONDARY OUTCOMES:
Overall survival (OS) | 24 months
  OS is the length of time from the date of inclusion until death from any cause.
Objective response rate (ORR) | 12 months
  ORR, as determined based on tumor response according to RECIST 1.1, is defined as the proportion of all included patients whose best overall response (BOR) is either a complete response or partial response.
Adverse events | 24 months
  Safety will be evaluated according to the NCI CTCAE Version 4.03. All observations

CONTACTS AND LOCATIONS:
Overall Officials: Feng duan, MD, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No